CLINICAL TRIAL: NCT05848076
Title: Effects of Therapeutic Neuroscience Education on Nociplastic Pain and Disability in Patients With Chronic Low Back Pain
Brief Title: Effects of Therapeutic Neuroscience Education in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AH/23/0105/ume Habiba
Record Dates: First submitted 2023-04-18; First posted 2023-05-08 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Chronic Low-back Pain
Keywords: back pain; therapuetic neuroscience education; range of motion
MeSH Terms: conditions — Back Pain | interventions — Core Stability

STUDY DESIGN:
Intervention Model Description: blinding
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNE with core stability (Experimental): Group A (TNE WITH CORE STABILITY) on low back this McGill exercise focuses on the ability of the spine to stabilize in different positions 3 sets of 3 repletion with of each of muscle and briefly explain the patient about their pain.The study participants will receive the total 18 session over 6 weeks period consider 3 treatment session per week
  Interventions: Other: TNE; Other: core stability
- Core stability (Active Comparator): McGill exercises for the low back. involved 3 sets of 3 repetitions for each muscle with a 30-second hold and 30-second rest interval for each repetition. The researcher will reassess the patient. Post treatment patient will complete Numeric Pain Rating Scale (NPRs), range of motion (Goniometer and Oswestry disability index (ODI). All study participant will receive a total of 18 treatment sessions over a six-week period, which consisted of 03 treatment sessions per week.
  Interventions: Other: core stability

INTERVENTIONS:
Other: TNE — McGill exercise focuses on the ability of the spine to stabilize in different positions 3 sets of 3 repletion with of each of muscle and briefly explains the patient about their pain
  Arms: TNE with core stability
Other: core stability — McGill exercises for the low back.

SUMMARY:
The study will be Randomized controlled trail, Subject diagnosed with low back pain meeting predetermined inclusion and exclusion criteria will be divided into two groups.

Pre assessment will be done using pain and disability as subjective measurement through Numeric pain rating scale (NPRS) & modified Oswestry disability index and the lumber range by goniometer as objective measurement. One group is subject will be treated with therapeutic neuroscience education and core stability exercise and second group is core stability exercise. Each subject received 18 sessions with 3 treatments per week. Post treatment values recorded after the session.After data collection from defined study setting,data will be entered and analyzed at Riphah International University,Lahore

DETAILED DESCRIPTION:
Chronic low back pain (LBP) is very common musculoskeletal disorders and leading causes of disability worldwide. Numerous epidemiological data show that 11%-84% of people experience, have experienced,or will experience pain in the lower spine at least once in their lives . With a global prevalence of 9.4%, LBP was ranked highest in the number of years lived with a disability and sixth in overall burden of disease Pakistan can suffer 56% from the LBP Nociplastic pain can be mechanistically defined as pain arising from the altered function of pain-related sensory pathways in the periphery and CNS, causing increased sensitivity Nociplastic pain should be viewed as an overarching terminology that can be applied to a diverse range of clinical conditions that share common neurophysiological mechanisms.

The main concern of TNE concept is that increasing the patient feeling of biology and physiology underpinning their pain condition instead of focus on anatomy and structure issues of tissue.In order to improve health of patient with CLBP healthcare provider proper educate their patient about experiencing pain and it may not result of tissue damage Several non surgical treatments have been offered to help and decrease LBP, such as joint manipulation, traditional therapeutic exercises , and medication

core stability training (CST) program this type of exercise focuses on the ability of the spine to stabilize in different positions and emphasize smaller, deeper, and posterior muscles. By increasing the endurance of these muscles, they retrain and maintain the correct physical condition to stabilize the spine to improve pain, performance, and ROM

There are few studies in literature which compare the TNE effect with core stability exercisein CLBP however there have been no studies which can compare TNE with nociplastic pain which effects on CLBP

ELIGIBILITY:
Inclusion Criteria:

* Diffused chronic low back pain
* Stop movement due to fear of increasing pain
* Anxiety and sleep problem with CLBP
* Symptoms duration most of days in 6 months
* No treatment other than analgesics

Exclusion Criteria:

* Diabetes mellites
* Radiating pain
* Spine surgery, fracture, arthritis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale for pain | 3 weeks
  NPRS (numeric pain rating scale) NPRS is based on 11 points numerical rating scale for determining pain intensity, 0( no
  ;pain), 10 (worst pain imaginable) pain intensity
Modified Oswestry Disability index (Disability and function) | 3 weeks
  Modified Oswestry Disability index Urdu version of Modified Oswestry Disability Index has become one of the principal condition-specific outcome measures used in the management of spinal disorders. At the baseline assessment, following each exercise session during the 12-week intervention, and finally at the end of the intervention programme, the MODI scores will be recorded

SECONDARY OUTCOMES:
Goniometer (Range of Motion) | 3 weeks
  A goniometer is an instrument that measures the available range of motion at a joint. The art and science of measuring the joint ranges in each plane of the joint are called goniometry. To measure the range of motion physical therapists most commonly use a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal Investigator; Ume Habiba, Principal Investigator — Study Principle Investigator
Locations (1):
- District Headquarter Hospital Layyah, Layyah, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No